CLINICAL TRIAL: NCT01751451
Title: A Phase 2, Randomized, 3-arm Study of Abiraterone Acetate Alone, Abiraterone Acetate Plus Degarelix, a GnRH Antagonist, and Degarelix Alone for Patients With Prostate Cancer With a Rising PSA or a Rising PSA and Nodal Disease Following Definitive Radical Prostatectomy
Brief Title: 3-arm Study of Abiraterone Acetate Alone, Abiraterone Acetate Plus Degarelix, a GnRH Antagonist, and Degarelix Alone for Patients With Prostate Cancer With a Rising PSA or a Rising PSA and Nodal Disease Following Definitive Radical Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); OHSU Knight Cancer Institute (Other); Rutgers Cancer Institute of New Jersey (Other); Endeavor Health (Other); Duke University (Other); Northwestern University Feinberg School of Medicine (Other); Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other); University of North Carolina (Other); Wayne State University (Other); Perlmutter New York University Cancer Center (Other); Weill Medical College of Cornell University (Other); Ferring Pharmaceuticals (Industry); GU Research Network, LLC (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-187
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Results first posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer
Keywords: ABIRATERONE ACETATE (CB 7630); DEGARELIX; PREDNISONE; 12-187
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

ARMS (3):
- Abiraterone acetate (Experimental): Group 1
  * Abiraterone acetate 1000 mg daily x 8 months
  * Prednisone 5 mg once daily x 8 months
  Interventions: Drug: Abiraterone acetate
- Abiraterone acetate and Degarelix (Experimental): Group 2
  Abiraterone acetate 1000 mg daily x 8 months
  * Prednisone 5 mg once daily x 8 months
  * Degarelix subcutaneous depot injection q 1 month x 8 months
  Interventions: Drug: Abiraterone acetate plus degarelix
- Degarelix (Experimental): Group 3
  • Degarelix subcutaneous depot injection q 1 month x 8 months
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Abiraterone acetate — Patients randomized to abiraterone acetate and prednisone (Group 1) will be instructed to take 1000 mg (four 250 mg tablets) of abiraterone acetate orally (PO) at least 1 hour before a meal and 2 hours after a meal every day. These patients will also be treated with prednisone 5 mg once daily with food.
  Arms: Abiraterone acetate
Drug: Abiraterone acetate plus degarelix — Patients randomized to abiraterone acetate plus degarelix and prednisone (Group 2) will be instructed to take 1000 mg (four 250 mg tablets) of abiraterone acetate orally (PO) at least 1 hour before a meal and 2 hours after a meal every day and prednisone 5 mg once daily with food. Patients will also be given two subcutaneous injections of degarelix 120 mg on Cycle 1, Day 1(starting dose) and 80 mg subcutaneous doses (maintenance doses) every 28 days (±3 days) thereafter.
  Arms: Abiraterone acetate and Degarelix
Drug: Degarelix — Patients randomized to degarelix alone (Group 3) will be given two subcutaneous injections of degarelix 120 mg on Cycle 1, Day 1 (starting dose) and 80 mg subcutaneous doses (maintenance doses) every 28 days (± 3 days) thereafter.
  Arms: Degarelix

SUMMARY:
In April 2011, the United States Food and Drug Administration (FDA) approved the oral drug abiraterone acetate (Zytiga ®) in combination with prednisone (a steroid) to treat patients with metastatic castration-resistant prostate cancer who have received prior docetaxel (chemotherapy). In December 2012, the FDA approved Zytiga ® in combination with prednisone to treat patients with metastatic castration-resistant prostate cancer who have not received prior chemotherapy. Degarelix (Firmagon ®), a testosterone lowering agent given as a monthly injection, is FDA approved for the treatment of patients with advanced prostate cancer. The purpose of this study is to evaluate abiraterone acetate and prednisone in combination with degarelix as a possible treatment for PSA recurrent prostate cancer as compared to abiraterone acetate alone and degarelix alone. This will be the first time these drugs will be used together.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent and Authorization for Use and Release of Health and Research Study Information (HIPAA authorization) NOTE: HIPAA authorization may be either included in the informed consent or obtained separately.
* Male aged 18 years and above
* Patients must have undergone local treatment via radical prostatectomy
* Patients who have received primary radiation therapy followed by a salvage radical prostatectomy are eligible.
* Patients who have had post-operative radiation therapy for presumed locally recurrent disease are eligible
* Histologically confirmed prostate cancer (per standards at Institution of participant registration) currently with progressive disease, defined as:
* Rising PSA (50% or more increase to a level of 1 ng/mL or more, based on at least 3 PSA determinations obtained at least 1 week apart). The 50% rise in PSA is across the 3 determinations, and these determinations do not need to be sequential AND
* PSADT ≤ 9 months as calculated according to the Memorial Sloan-Kettering Cancer Center nomogram (http://www.mskcc.org/mskcc/html/10088.cfm) OR
* Rising PSA as defined above AND
* Metastatic disease limited to the presence of pelvic and/or retroperitoneal nodes < 2 cm in short axis.
* Patients must have a serum testosterone of 150 ng/dL or greater
* ECOG performance status of ≤ 2 (Appendix A)
* Adequate bone marrow, hepatic, and renal function, as evidenced within 14 days prior to treatment initiation by:
* Absolute neutrophil count (ANC) ≥ 1500/mm3
* Platelet count ≥ 100,000/mm3
* Hemoglobin ≥ 9 g/dL without need for hematopoietic growth factor or transfusion support within 30 days prior to treatment initiation
* Aspartate aminotransferase (AST) ≤ 1.5 times the upper limit of the normal range (x ULN)
* Alanine aminotransferase (ALT) ≤ 1.5 x ULN
* Total bilirubin ≤ 1.5 x ULN
* Serum creatinine of ≤ 1.5 mg/dl or Calculated creatinine clearance of ≥ 60 mL/min
* Serum albumin ≥ 3.0 g/dL
* Serum potassium ≥ 3.5 mEq/L
* Prothrombin time (PT) ≤ 1.5 x ULN (or international normalized ratio [INR] ≤ 1.3) unless the patient is receiving anticoagulant therapy
* Partial thromboplastin time (PTT) ≤ 1.5 x ULN unless the patient is receiving anticoagulant therapy At least 4 weeks and recovery to Grade 0-1 from reversible effects of prior surgery (i.e., incisional pain, wound drainage)
* Able to swallow the study drug whole as a tablet
* Willing to take abiraterone acetate on an empty stomach; no food should be consumed at least two hours before and for at least one hour after the dose of abiraterone acetate is taken
* Patients who have partners of childbearing potential must be willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator during the study and for 1 week after last dose of abiraterone acetate.

Exclusion Criteria:

* Prior cytotoxic chemotherapy or biologic therapy for prostate cancer
* More than 8 months of prior hormonal therapy (e.g., gonadotropin-releasing hormone analogs, megestrol acetate, or Casodex) Note: Patients who have been on prior hormonal therapy must wait at least 1 year after the drug is fully metabolized to start treatment on protocol.
* Prior ketoconazole, abiraterone acetate, or enzalutamide for the treatment of prostate cancer.
* Known brain metastasis or evidence of metastatic disease by CT scan, physical exam, or bone scan within 4 weeks of registration
* Patients with equivocal uptake on a bone scan that in the clinician's opinion do not definitively constitute metastatic disease are eligible
* Currently active second malignancy

Significant medical condition other than cancer, that would prevent consistent and compliant participation in the study that would, in the opinion of the investigator, make this protocol unreasonably hazardous including but not limited to:

* Active infection or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated
* Severe hepatic impairment (Child-Pugh Class C)
* History of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of the study agents
* Uncontrolled hypertension (systolic BP ≥ 160 mmHg or diastolic BP ≥ 95 mmHg); patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment
* Active or symptomatic viral hepatitis or chronic liver disease
* History of pituitary or adrenal dysfunction
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class III or IV heart disease or cardiac ejection fraction measurement of < 50 % at baseline
* Atrial fibrillation, or other cardiac arrhythmia requiring medical therapy
* Uncontrolled diabetes mellitus
* Active psychiatric condition Use of any prohibited concomitant medications (Section 5.5) within 30 days prior to Cycle 1, Day 1
* Pre-existing condition that warrants long-term corticosteroid use in excess of study dose
* Grade > 2 treatment-related toxicity from prior therapy
* Known allergies, hypersensitivity or intolerance to abiraterone acetate, prednisone or degarelix
* Administration of an investigational therapeutic within 30 days of Cycle 1, Day1
* Any condition which, in the opinion of the investigator, would preclude participation in this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2012-12-18 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard I Scher, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (16):
- United States (16):
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Karmanos Cancer Institute, Wayne State University, Detroit, Michigan
  - Urology Cancer Center and GU Research Network, Omaha, Nebraska
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - NorthShore University Health System, Long Island City, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center at Phelps, Sleepy Hollow, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health & Science University Knight Cancer Institute, Portland, Oregon

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Abiraterone Acetate: Group 1
  * Abiraterone acetate 1000 mg daily x 8 months
  * Prednisone 5 mg once daily x 8 months
  Abiraterone acetate: Patients randomized to abiraterone acetate and prednisone (Group 1) will be instructed to take 1000 mg (four 250 mg tablets) of abiraterone acetate orally (PO) at least 1 hour before a meal and 2 hours after a meal every day. These patients will also be treated with prednisone 5 mg once daily with food.
- Abiraterone Acetate and Degarelix: Group 2
  Abiraterone acetate 1000 mg daily x 8 months
  * Prednisone 5 mg once daily x 8 months
  * Degarelix subcutaneous depot injection q 1 month x 8 months
  Abiraterone acetate plus degarelix: Patients randomized to abiraterone acetate plus degarelix and prednisone (Group 2) will be instructed to take 1000 mg (four 250 mg tablets) of abiraterone acetate orally (PO) at least 1 hour before a meal and 2 hours after a meal every day and prednisone 5 mg once daily with food. Patients will also be given two subcutaneous injections of degarelix 120 mg on Cycle 1, Day 1(starting dose) and 80 mg subcutaneous doses (maintenance doses) every 28 days (±3 days) thereafter.
- Degarelix: Group 3
  • Degarelix subcutaneous depot injection q 1 month x 8 months
  Degarelix: Patients randomized to degarelix alone (Group 3) will be given two subcutaneous injections of degarelix 120 mg on Cycle 1, Day 1 (starting dose) and 80 mg subcutaneous doses (maintenance doses) every 28 days (± 3 days) thereafter.
Period: Overall Study
Arm/Group | Abiraterone Acetate | Abiraterone Acetate and Degarelix | Degarelix
Started | 42 | 40 | 42
Completed | 42 | 40 | 42
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abiraterone Acetate | Abiraterone Acetate and Degarelix | Degarelix | Total
Number analyzed (Participants) | 42 | 40 | 42 | 124
Age, Continuous [Mean (Full Range); unit: years] | 63.6 [43 to 83] | 66.2 [55 to 81] | 63.7 [20 to 78] | 64.5 [20 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 42 | 40 | 42 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 42 | 40 | 41 | 123
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 3 | 11
  White | 37 | 31 | 38 | 106
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 5 | 1 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 40 | 42 | 124

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: defined as an undetectable PSA (using a routine non-ultrasensitive PSA assay) with non-castrate level of testosterone (>150 ng/dL) at 18 months from the time of treatment initiation (PSA0).
Time Frame: 18 months
Measure: Mean (95% Confidence Interval); unit: percentage change of PSA
Arm/Group | Abiraterone Acetate | Abiraterone Acetate and Degarelix | Degarelix
Number analyzed (Participants) | 42 | 40 | 42
percentage change of PSA | 5.1 [1 to 17] | 17.1 [7 to 32] | 11.9 [4 to 26]

2. Primary Outcome: Soft Tissue Complete Response
Description: In addition to an undetectable PSA, any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm (Complete Response per RECIST) in order to meet the criteria for PFS. Outcome in subjects who develop radiographically evident metastatic disease while on study will be considered treatment failures independent of their respective PSA values.
Time Frame: 1 year
Population: N/A - data were not collected
Arm/Group | Abiraterone Acetate | Abiraterone Acetate and Degarelix | Degarelix
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: PSA Response Rate
Description: The percentage of patients with a non-castrate level of testosterone (>150 ng/dL) and an undetectable PSA at 8 months from PSA0 will be measured.
Time Frame: 8 months
Population: N/A - data were not collected
Arm/Group | Abiraterone Acetate | Abiraterone Acetate and Degarelix | Degarelix
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Overall Quality of Life
Description: with particular attention to libido, potency, anxiety, depression, hot flashes, and fatigue. Effects of each arm on health-related quality of life will be assessed via PRO Survey (Appendix C) completed on paper by the patient at the following study visits: Up to 30 Days Prior to Randomization, each Day 1 of Treatment Cycle, End of Treatment, and each Post-Treatment Follow-up.Effects of each arm on quality of life,
Time Frame: 1 year
Population: N/A - data were not collected
Arm/Group | Abiraterone Acetate | Abiraterone Acetate and Degarelix | Degarelix
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Non-hematologic Adverse Events
Description: Safety will be evaluated according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Safety assessments will be based on medical review of adverse event reports and the results of vital sign measurements, physical examinations and clinical laboratory tests throughout the conduct of the study.
Time Frame: 1 year
Population: N/A - data were not collected
Arm/Group | Abiraterone Acetate | Abiraterone Acetate and Degarelix | Degarelix
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Testosterone and Luteinizing Hormone (LH) Recovery Rates
Description: Testosterone and LH recovery rates will be measured at 8 months from the start of randomization and at each month of the 10 month follow up period.
Time Frame: 8 -10 months
Population: N/A - data were not collected
Arm/Group | Abiraterone Acetate | Abiraterone Acetate and Degarelix | Degarelix
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Correlative Tissue Analysis
Description: Tissue samples will be utilized for morphologic assessment, percent tumor involvement (if applicable), and immunohistochemistry. The immunohistochemical markers assessed may be AR, PTEN, PSMA, fatty acid synthase (FASN), phospho-AMPK, phospho-ACC, phospho-S6 kinase, phospho-Akt for the assessment of the AMPK, lipid synthesis, mTOR pathways, and immunological markers.
Time Frame: 1 year
Population: N/A - data were not collected
Arm/Group | Abiraterone Acetate | Abiraterone Acetate and Degarelix | Degarelix
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Abiraterone Acetate | Abiraterone Acetate and Degarelix | Degarelix
All-Cause Mortality (participants affected / at risk) | 2/42 | 3/40 | 0/42
Serious Adverse Events (participants affected / at risk) | 2/42 | 5/40 | 4/42
Other Adverse Events (participants affected / at risk) | 5/42 | 5/40 | 4/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate (N=42) | Abiraterone Acetate and Degarelix (N=40) | Degarelix (N=42)
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1
Aortic valve disease (Cardiac disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fever (General disorders) | 2 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pelvic infection (Infections and infestations) | 1 | 0 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 0 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Stroke (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate (N=42) | Abiraterone Acetate and Degarelix (N=40) | Degarelix (N=42)
Alanine aminotransferase increased (Investigations) | 1 | 3 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 2 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT01751451/Prot_SAP_000.pdf